CLINICAL TRIAL: NCT04343703
Title: Suicide Prevention and Intervention (SURVIVE): Cohort Study and Nested Randomized Controlled Trials of Secondary Prevention Programs for Suicide Attempts
Brief Title: Suicide Prevention and Intervention in Spain: the SURVIVE Study
Acronym: SURVIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Víctor Pérez, Medical Director, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/8629/I
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Suicide; Suicide, Attempted; Depression
Keywords: suicide; suicide attempted; depression; secondary prevention; mental health
MeSH Terms: conditions — Suicide; Suicide, Attempted; Depression; Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Telephone-based management (Experimental): Telephone-based management will consist of a three-phase intervention: 1) An initial 15-20 min call at 1 week of enrollment in which the cases manager introduces him/herself, and does a short assessment of the current suicide risk, 2) A 5-10 min telephone follow-up at 1, 3, 6, 9 and 12 months, 3) If suicide risk is detected, a 15-45 min crisis intervention call will be done, tailored to the participant's characteristics and context. If deemed necessary, an emergency face-to-face appointment will be scheduled. At each phone call information regarding the current treatment, adherence to mental health services, and current life stressors will be collected.
  Interventions: Behavioral: Treatment as Usual
- iFightDepression for Suicide (Experimental): The iFightDepression-Survive (iFD-S) program is a cognitive-behavioral, internet-based self-management tool, developed by the European Alliance Against Depression (EAAD). The iFD is intended to address mild-to-moderate depressive symptoms. The iFD tool is structured in seven core modules focused on: behavioral activation, cognitive restructuring, sleep regulation, mood monitoring, and healthy lifestyle habits. The content of each module is intended to be followed over 1 week and consists of written information, tasks to do over the week and worksheets. All of these aims to consolidate learning and promote self-monitoring. For this study, an additional module (iFD-S) will be developed. To that end, the expertise of a panel of mental health experts in suicide and cognitive-behavioral interventions will be asked. The iFD-S also provides telephone guidance (2h per participant) during the use of the program.
  Interventions: Behavioral: Treatment as Usual
- Treatment as Usual (Active Comparator): Treatment as Usual (TaU) will vary across sites, however it generally implies a combination of case management strategies (including telephone calls, visits by mental health services) and pharmacotherapy. For this study, any nonspecific intervention to address suicidal behavior or to prevent suicide will be considered as treatment as usual. TaU will consist of any routine procedures applied at each participating site.
  Interventions: Behavioral: Telephone-based management; Behavioral: iFightDepression for Suicide
- Self Awareness of Mental Health (Experimental): The Self Awareness of Mental Health (SAM) is an adaptation of the Youth Awareness of Mental Health program, originally developed for the Saving and Empowering Young Lives in Europe (SEYLE) study. The SAM aims to raise mental health awareness about risk and protective factors associated with suicide, provide knowledge about depression and anxiety, and enhance the skills needed to cope with adverse life events and suicidal behavior. The intervention is delivered by trained clinical psychologists in five, 45-60 minutes, face-to-face sessions.
  Interventions: Behavioral: Treatment as Usual; Behavioral: Self Awareness of Mental Health

INTERVENTIONS:
Behavioral: Telephone-based management — The intervention consists of a series of phone calls aimed at providing follow up care of individuals at risk. At each phone call the case manager collects information regarding the current treatment, adherence to mental health services, and current life stressors.
  Arms: Treatment as Usual
Behavioral: iFightDepression for Suicide — The iFD-Survive is a cognitive-behavioral, internet-based self-management tool, developed by the European Alliance Against Depression (EAAD). The iFD is intended to address mild-to-moderate depressive symptoms. The iDF tool is structured in seven core modules focused on: behavioral activation, cognitive restructuring, sleep regulation, mood monitoring, and healthy lifestyle habits. The content of each module is intended to be followed over 1 week and consists of written information, tasks to do over the week and worksheets. All of these aims to consolidate learning and promote self-monitoring. For this study, an additional module (iFD-S) will be developed. The iFD-S also provides telephone guidance (2h per participant).
  Other Names: iFD-S
  Arms: Treatment as Usual
Behavioral: Treatment as Usual — Treatment as Usual (TaU) will vary across sites, however it generally implies a combination of case management strategies (including telephone calls, visits by mental health services) and pharmacotherapy. For this study, any nonspecific intervention to address suicidal behavior or to prevent suicide will be considered as treatment as usual.
  Other Names: TaU
  Arms: Self Awareness of Mental Health; Telephone-based management; iFightDepression for Suicide
Behavioral: Self Awareness of Mental Health — The SAM consist of five, face-to-face, individual sessions designed to raise awareness about depression, anxiety and suicidal behaviors as well as to enhancing skills to effectively cope with stressful life events and mood.
  Other Names: SAM
  Arms: Self Awareness of Mental Health

SUMMARY:
Suicide is one of the leading causes of avoidable death worldwide. Gathering population-representative data on the incidence of suicidal behavior, as well as developing effective secondary prevention strategies are imperative parts of evidence-based public health policies, currently lacking in Spain. The Suicide Prevention and Intervention Study (SURVIVE) is a multi-site-cohort study with nested randomized-controlled clinical trials. The principal aims of the SURVIVE study are to determine the incidence of suicide attempts in Spain and to investigate the efficacy of two secondary prevention programs.

DETAILED DESCRIPTION:
Suicide is the leading cause of avoidable death worldwide, demanding urgent attention. Collecting national-representative data is the first step towards developing effective evidence-based public-policies.

The SURVIVE study presents four inter-connected objectives:

1. To determine the incidence of suicide attempts in Spain
2. To follow up suicide attempters with the aim of studying the probability of them re-attempting
3. To identify influential risk factors to explain suicide attempts and an increased risk of re-attempting
4. To determine the efficacy of secondary prevention programs to prevent suicide re-attempts in comparison to treatment as usual (TAU).

Study design: Multi-site-coordinated cohort study with nested randomized controlled trials. Participants will be recruited at mental-health sites distributed across Spain.

Participants: A cohort of 2.000 individuals presenting a suicide attempt will be established.

Individuals would be followed for 1-year, and assessed every 3 months.

Participants (age >18) that meet inclusion/exclusion criteria will be randomly allocated to:

1) telephone-based management, or 2) iFightDepression for Suicide (iFD-Survive), a web-based-self-management tool. These interventions will be tested against TAU.

Participants (age between 12-17) that meet inclusion/exclusion criteria will be randomly allocated to: 1)a face-to-face individual intervention designed for youths Specific Aware of Mental Health Intervention for adolescents (SAM) or 2) TAU.

ELIGIBILITY:
General Inclusion Criteria:

* Female and males, age >= 12 years
* Having attended a hospital emergency department due to a suicide attempt
* Willing and able to comply with study procedures and to give written informed consent

Specific inclusion criteria for iFD-S:

* Minimum knowledge of internet use and availability of an internet device (tablet, computer, smartphone)
* Depressive symptoms according to PHQ-9 scores above 15

Specific inclusion criteria for SAM:

* Age between 12-17
* Informed consent of legal guardians

General Exclusion Criteria:

* Incapacity to give informed consent
* Lack of fluency in Spanish
* Currently taking part in another clinical study which, in the opinion of the investigator, is likely to interfere with the objectives of the SURVIVE study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1742 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Suicide repetition (or death by suicide) | 12 months
  The primary outcome is subsequent suicide attempts (and/or suicide mortality) captured across assessment points. Is a binary variable (yes/no).

SECONDARY OUTCOMES:
Brief Symptoms Inventory | 1 month
  The BSI is a 53-item self-report scale designed to evaluate psychopathological and psychological symptoms, measuring nine dimensions (i.e.,somatization, obsession-compulsion, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism) that can be summed up to reflect three global indices. These synthetic indices are the General Severity Index (GSI), the Positive Symptom Distress Index, and the Positive Symptom Total. In more detail, the BSI uses a 5-point Likert scale, ranging from 0 ("not at all") to 4 ("extremely"). Scores range from 0 to 212, higher scores mean a worse outcome.
Patient Health Questionnaire 9-items | 2 weeks
  The PHQ-9 measures depressive symptoms in a scale from 0 (not at all) to 3 (nearly every day). Scores range from 0 to 27 and higher scores mean a worse outcome. The PHQ-9 A will be used for participants aged 12-17.
Generalized Anxiety Disorder 7-items | 2 weeks
  GAD-7 consists of seven items measuring worry and anxiety symptoms. Each item is scored on a four-point Likert scale (0-3) with total scores ranging from 0 to 21 with higher scores reflecting greater anxiety severity.
EuroQol 5D | 1 day
  Part one provides a self-reported description of health problems into five dimensions. Patients have to rate the severity of each dimension in a 5-point scale. For part one, higher scores represent a worse outcome (less quality of life).Part two consist of a Visual Analogue Scale corresponding to the current state of the subject's health. The lowest extreme (0) corresponds to the worst imaginable state, and the highest extreme (100) represents the best imaginable health state.
Barrat Impulsivity Scale | 2 weeks
  The BIS is a 30-item widely used questionnaire that measures three aspects of impulsivity: 1) motor impulsiveness (acting without forethought), 2) attentional impulsiveness (tendency to make quick, non-reflexive decisions), and 3) non-planned impulsiveness (failure to prepare for future events). Each item is rated in a 4 point scale (0-4). Total scores range from 0 to 44, higher scores represent higher impulsivity.
Acquired capability of suicide Scale -Fearlesness about Death | 2 weeks
  Acquired Capability for Suicide Scale-Fearlessness about Death (ACSS-FAD) is a seven-item self-report measure which uses a 5-point Likert scale ranging from 0 (not at all like me) to 4 (very much like me). Scores range from 0 to 32, and higher scores represent a worse outcome (higher levels of the acquired capability for suicide).
Reflective Functioning Questionnaire | 2 weeks
  The 8-item version of the Reflective Functioning Questionnaire is a self-reported instrument that measures reflective functioning, an expression of mentalizing processes. The instrument separately addresses the levels of both certainty and uncertainty about one's own mental processes. Items are scored in a 7 point-scale (1 to 7), meaning that the total score ranges from 8 to 56, higher scores represent a higher capacity of mentalizing, and therefore a better outcome.
Columbia Suicide Rating Scale | 1 month
  The Columbia Suicide Rating Scale is a suicidal ideation and behavior rating scale that evaluates suicide risk.It rates an individual's degree of suicidal ideation on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent and behaviors. It contains 6 "yes" or "no" questions in which respondents are asked to indicate whether they have experienced several thoughts or feelings relating to suicide over the past month and behaviors over their lifetime and past 3 months. An answer of "yes" to any of the six questions may indicate a need for referral and an answer of "yes" to questions 4, 5 or 6 indicate high-risk.
Strengths and Difficulties Questionnaire (SDQ) | 1 month
  Emotional and behavioral screening questionnaire designed for youths.

CONTACTS AND LOCATIONS:
Overall Officials: Víctor Pérez, PhD, Principal Investigator — Parc de Salut Mar
Locations (8):
- Spain (8):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Santiago de Áraba, Vitoria-Gasteiz, Basque Country
  - Institute of Neuropsychiatry and Addictions, INAD, Parc de Salut Mar, Barcelona, Catalonia
  - Hospital Clinic, Barcelona, Catalonia
  - Corporació Sanitaria Parc Tauli, Sabadell, Catalonia
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Perez V, Elices M, Toll A, Bobes J, Lopez-Sola C, Diaz-Marsa M, Grande I, Lopez-Pena P, Rodriguez-Vega B, Ruiz-Veguilla M, de la Torre-Luque A; SURVIVE Group. The Suicide Prevention and Intervention Study (SURVIVE): Study protocol for a multisite cohort study with nested randomized-controlled trials. Span J Psychiatry Ment Health. 2023 Jan-Mar;16(1):16-23. doi: 10.1016/j.rpsm.2020.11.004. Epub 2020 Dec 7. PMID 33301997